CLINICAL TRIAL: NCT07085767
Title: A Phase 3 Randomized, Double-Blind, Active-Controlled Study of Palazestrant With Ribociclib Versus Letrozole With Ribociclib for the First-Line Treatment of ER+, HER2- Advanced Breast Cancer (OPERA-02)
Brief Title: Palazestrant in Combination With Ribociclib for the First-line Treatment of ER+/HER2- Advanced Breast Cancer
Acronym: OPERA-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Olema Pharmaceuticals, Inc. (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OP-1250-302; OPERA-02 (Other: Olema Pharmaceuticals, Inc.)
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Locally Advanced Breast Cancer; Metastatic Breast Cancer; ER Positive Breast Cancer; HER2 Negative Breast Carcinoma
Keywords: Randomized; Multicenter; Double-Blind; Active-Controlled; Phase 3; Palazestrant; Complete Estrogen Receptor Antagonist (CERAN); Selective Estrogen Receptor Degrader (SERD); Ribociclib; CDK4/6i; Letrozole; Aromatase inhibitors; Antineoplastic agents
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Palazestrant (Experimental): Participants will receive palazestrant, ribociclib and letrozole-matching placebo
  Interventions: Drug: Palazestrant; Drug: Letrozole-matching placebo; Drug: Ribociclib
- Letrozole (Active Comparator): Participants will receive letrozole, ribociclib and palazestrant-matching placebo
  Interventions: Drug: Ribociclib; Drug: Letrozole; Drug: Palazestrant matching-placebo

INTERVENTIONS:
Drug: Palazestrant — Participants will be treated with palazestrant 90 mg once daily on a 4-week (28-day) cycle.
  Other Names: OP-1250
  Arms: Palazestrant
Drug: Letrozole-matching placebo — Participants will be treated with letrozole-matching placebo once daily on a 4-week (28 day) cycle
  Arms: Palazestrant
Drug: Ribociclib — Participants will be treated with ribociclib 600 mg once daily on Days 1-21 of a 4-week (28 day) cycle.
Drug: Letrozole — Participants will be treated with letrozole 2.5 mg once daily on a 4-week (28-day) cycle
  Arms: Letrozole
Drug: Palazestrant matching-placebo — Participants will be treated with palazestrant-matching placebo once daily on a 4-week (28-day) cycle
  Arms: Letrozole

SUMMARY:
This phase 3 clinical trial compares the efficacy and safety of palazestrant with ribociclib to letrozole and ribociclib in women and men who have not received prior systemic anti-cancer treatment for advanced breast cancer.

DETAILED DESCRIPTION:
This is an international, multicenter, randomized, double-blind, active-controlled, phase 3 clinical trial. The purpose of this trial is to compare the efficacy and safety of palazestrant in combination with ribociclib +letrozole -matching placebo (Arm A: investigational arm) with letrozole in combination with ribociclib + palazestrant-matching placebo (Arm B: control arm).

This trial is seeking adult participants with ER+, HER2- advanced breast cancer who have not received prior systemic anti-cancer treatment for advanced disease. Approximately 1,000 participants will be randomized in a 1:1 ratio to one of the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Adult female or male participants.
* ER+, HER2- locally advanced or metastatic breast cancer that is not amenable to curative therapy.
* Evaluable disease (measurable disease per RECIST 1.1 or bone-only disease).
* De novo advanced breast cancer or with disease recurrence occurring after 12 months of completing adjuvant endocrine therapy (with or without CDK4/6 inhibitors)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, hepatic, and renal functions.
* Female participants can be pre-, peri- or postmenopausal.
* Male and pre- or peri-menopausal female participants must be willing to take a GnRH (or LHRH) agonist.

Exclusion Criteria:

* Disease recurrence during adjuvant endocrine therapy
* Currently receiving or previously received systemic anti-cancer therapy for ER+, HER2- advanced breast cancer.
* Previously received treatment with fulvestrant, elacestrant or an investigational endocrine therapy in any setting.
* History of allergic reactions to study treatment.
* Any contraindications to letrozole and ribociclib.
* Symptomatic central nervous system metastases, carcinomatous meningitis, leptomeningeal disease, or a spinal cord compression that require immediate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From Date of Randomization until Disease Progression or Death Due to Any Cause (estimated as up to 3.5 years)
  To compare PFS, based on a local investigator assessment, between investigational (palazestrant with ribociclib + letrozole-matching placebo) and control (letrozole with ribociclib + palazestrant-matching placebo) arms.

SECONDARY OUTCOMES:
Overall Survival (OS) | From Date of Randomization until Death Due to Any Cause (estimated as up to 5.5 years)
  To compare OS between investigational and control arms.
Progression Free Survival (PFS) | From Date of Randomization until Disease Progression or Death Due to Any Cause (estimated as up to 3.5 years)
  To evaluate PFS based on Blinded Independent Review Committee (BIRC) assessment
Overall response Rate (ORR) | From Date of Randomization until Tumor Response (estimated as up to 3.5 years)
  To evaluate ORR based on Blinded Independent Review Committee (BIRC) assessment
Duration of Response (DOR) | From Date of Tumor Response (CR or PR) until Disease Progression (estimated as up to 3.5 years)
  To evaluate DOR based on Blinded Independent Review Committee (BIRC) assessment
Clinical Benefit Rate (CBR) | Proportion of subjects achieving CR, PR or SD with duration of at least 24 weeks (estimated as up to 3.5 years)
  To evaluate CBR based on Blinded Independent Review Committee (BIRC) assessment
Overall response Rate (ORR) | From Date of Randomization until Tumor Response (estimated as up to 3.5 years)
  To evaluate ORR based on local investigator assessment
Duration of Response (DOR) | From Date of Tumor Response (CR or PR) until Disease Progression (estimated as up to 3.5 years)
  To evaluate DOR based on local investigator assessment
Clinical Benefit Rate (CBR) | Proportion of subjects achieving CR, PR or SD with duration of at least 24 weeks (estimated as up to 3.5 years)
  To evaluate CBR based on local investigator assessment
Safety and tolerability | Up to 42 days after end of treatment (estimated as up to 3.5 years)
  To evaluate safety and tolerability assessed by AEs, SAEs, dose modifications, clinical laboratory parameters, ECGs, performance status and vital sign measurements
Pharmacokinetics (PK) of palazestrant and ribociclib | Every 28 days (estimated as up to 3.5 years)
  To evaluate plasma levels of palazestrant and ribociclib to establish pharmacokinetic (PK) parameters
Health-related patient-reported outcomes (PROs) | Every 28 days (estimated as up to 3.5 years)
  To evaluate the change from baseline in health-related PROs assessed using standardized instruments that are widely used in (breast) cancer clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Olema Pharmaceuticals, Inc.
Locations (22):
- United States (8):
  - Clinical Trial Site, Ames, Iowa
  - Clinical Trial Site, Scarborough, Maine
  - Clinical Trial Site, Kansas City, Missouri
  - Clinical Trial Site, Santa Fe, New Mexico
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Sayre, Pennsylvania
  - Clinical Trial Site, Tennessee City, Tennessee
  - Clinical Trial Site, Salt Lake City, Utah
- Australia (7):
  - Clinical Trial Site, Sydney, New South Wales
  - Clinical Trial Site, Waratah, New South Wales
  - Clinical Trial Site, South Brisbane, Queensland
  - Clinical Trial Site, Adelaide, South Australia
  - Clinical Trial Site, Clayton, Victoria
  - Clinical Trial Site, Geelong, Victoria
  - Clinical Trial Site, Nedlands, Western Australia
- Hong Kong (2):
  - Clinical Trial Site, Hong Kong, Kowloon
  - Clinical Trial Site, Hong Kong, Pok Fu Lam
- Taiwan (2):
  - Clinical Trial Site, Kaohsiung City, Sanmin
  - Clinical Trial Site, Chang-hua
- Thailand (3):
  - Clinical Trial Site, Dusit, Bangkok
  - Clinical Trial Site, Ban Phaeo, Changwat Samut Sakhon
  - Clinical Trial Site, Hat Yai, Changwat Songkhla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Olema Publications — https://olema.com/science/publications